CLINICAL TRIAL: NCT05596318
Title: Efficacy of Digital Cognitive Behavior Therapy for Insomnia for the Prevention of Perinatal Depression
Brief Title: Perinatal Research on Improving Sleep and Mental Health
Acronym: PRISM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-35440
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Insomnia; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Digital cognitive behavior therapy for insomnia (CBT-I) (Experimental)
  Interventions: Device: Digital CBT-I
- Digital sleep hygiene education (SHE) (Active Comparator)
  Interventions: Device: Digital SHE

INTERVENTIONS:
Device: Digital CBT-I — The digital CBT-I program is called Sleepio (Big Health, Ltd). Digital CBT-I will be delivered by an animated therapist in six weekly sessions that are approximately 10-20 minutes each. Sessions can be accessed via website or app at a time that is convenient for the participant. Session content is based on standard, in-person CBT-I protocols, and includes sleep restriction, stimulus control, cognitive therapy, relaxation techniques, and sleep hygiene education. The program is interactive, automated, and tailored to participant progress. Additionally, participants will receive supplemental CBT-I content tailored for prenatal and postpartum insomnia.
  Other Names: Sleepio
  Arms: Digital cognitive behavior therapy for insomnia (CBT-I)
Device: Digital SHE — The digital SHE program was created by Big Health, Ltd and has a total of six sessions. The content for SHE includes education about sleep stages, sleep architecture, sleep cycles; education about importance of sleep for performance, mood, and health; recommendations for developing healthy sleep habits; recommendations for lifestyle factors that impact sleep; recommendations for creating a sleep-friendly bedroom.
  Arms: Digital sleep hygiene education (SHE)

SUMMARY:
The goal of this clinical trial is to compare two sleep programs in pregnant people with insomnia. The main questions it aims to answer are:

1. What is the efficacy of digital cognitive behavioral therapy for insomnia (CBT-I) versus digital sleep hygiene education (SHE) for preventing perinatal depression?
2. Is the effect of digital CBT-I on perinatal depression mediated through prenatal insomnia symptom improvement?
3. Is the effect of digital CBT-I on perinatal depression moderated by baseline depressive symptom severity?

Participants will receive one of two sleep programs - SHE or CBT-I. Both involve six weekly online sessions. Participants will complete surveys and interviews until 1 year postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant 14-28 weeks gestation
* 18 years or older
* Daily access to a web-enabled computer, smart phone, or tablet
* Current elevated insomnia symptom severity and insomnia disorder
* English speaking

Exclusion Criteria:

* Current major depression
* Taking or planning to take antidepressant medication (ADM)
* Other diagnosed or suspected sleep disorder
* Other psychiatric or medical issues (e.g., bipolar disorder, active suicidality, bed rest)
* Night shift worker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of perinatal depression, as assessed by the Structured Clinical Interview for the DSM-5 (SCID) | Baseline to 12 months postpartum
  This is a binary outcome that measures whether a participant experienced a depressive episode at any point since randomization.

SECONDARY OUTCOMES:
Change in depressive symptom severity from baseline to 12 months postpartum, as assessed by the Edinburgh Postnatal Depression Scale (EPDS) | Baseline to 12 months postpartum
  The Edinburgh Postnatal Depression Scale (EPDS) score ranges from 0 to 30, with higher scores indicating greater depressive symptom severity.
Change in depressive symptom severity from baseline to 12 months postpartum, as assessed by the Patient Health Questionnaire-9 (PHQ-9) | Baseline to 12 months postpartum
  The Patient Health Questionnaire-9 (PHQ-9) score ranges from 0 to 27, with higher scores indicating greater depressive symptom severity.
Change in suicidal ideation severity, as rated by the C-SSRS | Baseline to 12 months postpartum
  The Columbia Suicide Severity Rating Scale suicidal ideation score ranges from 1-5, with greater scores indicating more severe ideation, based on the following categories:
  1. - Wish to be Dead
  2. - Non-specific Active Suicidal Thoughts
  3. - Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act
  4. - Active Suicidal Ideation with Some Intent to Act, without Specific Plan
  5. - Active Suicidal Ideation with Specific Plan and Intent
Change in anxiety symptom severity, as assessed by the GAD-7 | Baseline to 12 months postpartum
  The Generalized Anxiety Disorder-7 score ranges from 0 to 21, with higher scores indicating greater anxiety symptom severity.
Change in prenatal insomnia symptom severity as a mediator of the effect of digital CBT-I on perinatal depression, as assessed by the ISI | Baseline to 10 weeks post-randomization (mediator)
  The Insomnia Severity Index (ISI) score ranges from 0 to 28, with higher scores indicating greater insomnia severity.
Baseline depressive symptom severity as a moderator, as assessed by the EPDS | Baseline
  The Edinburgh Postnatal Depression Scale (EPDS) score ranges from 0 to 30, with higher scores indicating greater depressive symptom severity.
Baseline depressive symptom severity as a moderator, as assessed by the PHQ-9 | Baseline
  The Patient Health Questionnaire-9 (PHQ-9) score ranges from 0 to 27, with higher scores indicating greater depressive symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Felder, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data via the National Database for Clinical Trials related to Mental Illness (NDCT), which is a secure platform for scientific collaboration and data-sharing
Supporting Information: Study Protocol, SAP
Time Frame: Annually

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT05596318/Prot_SAP_000.pdf